CLINICAL TRIAL: NCT05613855
Title: Performance of Pulmonary Embolism Risk Scores for Assessment of Outcome in Computed Tomographic Pulmonary Angiography Confirmed Patients
Brief Title: Performance of Pulmonary Embolism Risk Scores Out Come in CTPA Confirmed Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nourhan Safwat Abdelraheem Hussien, Resident doctor, Assiut University
Other Study IDs: performance score outcome
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Assess performance of PERFORM score in predicting outcome in CTPA confirmed patients.
2. Compare PERFORM score with the currently validated PESI in risk stratification of patients

DETAILED DESCRIPTION:
Pulmonary embolism (PE) is a common and potentially lethal condition in the emergency department requiring early and accurate management.

The short-term mortality rate of PE varies widely and ranges from less than 2% in many patients with non massive PE to more than 95% in patients who experience cardiorespiratory arrest.

Although several prognostic models of acute PE are currently used, all of them have practical limitations.

Of all clinical scores integrating PE severity and comorbidity, the Pulmonary Embolism Severity Index (PESI) and its simplified version,(sPESI) have been most extensively validated to date.

However, current prognostic scores for pulmonary embolism (PE) are partly based on patients without PE confirmation via computed tomographic pulmonary angiography (CTPA), involving subjective parameters and complicated scoring methods [8].

Therefore, an objective, accurate, and simple prognostic model in CTPA-confirmed patients to predict the risk of 30-day mortality. help clinicians assess patients' risks and improve therapeutic decision-making that is called PERFORM score (pulmonary embolism risk score for mortality)

ELIGIBILITY:
Inclusion Criteria:

- Patients above 18 years old with PE confirmed by CTPA are considered for inclusion in the study.

Exclusion Criteria:

* • Patients who have contraindications for CTPA eg. Renal impairment

  * Patients diagnosed and treated as PE without doing CTPA.
  * Patients who refuse to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be on patients wh are above 18 years okd who are daignosed to have pulmonary embolism with CTPA
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Assess performance of PERFORM score in predicting outcome in CTPA confirmed patients. | from 11/2022 to 4/2024

SECONDARY OUTCOMES:
Compare PERFORM score with the currently validated PESI in risk stratification of patients. | from 11/2022 to 4/2024

REFERENCES:
- [Result] Anderson FA Jr, Wheeler HB, Goldberg RJ, Hosmer DW, Patwardhan NA, Jovanovic B, Forcier A, Dalen JE. A population-based perspective of the hospital incidence and case-fatality rates of deep vein thrombosis and pulmonary embolism. The Worcester DVT Study. Arch Intern Med. 1991 May;151(5):933-8. PMID 2025141
- [Result] Kurkciyan I, Meron G, Sterz F, Janata K, Domanovits H, Holzer M, Berzlanovich A, Bankl HC, Laggner AN. Pulmonary embolism as a cause of cardiac arrest: presentation and outcome. Arch Intern Med. 2000 May 22;160(10):1529-35. doi: 10.1001/archinte.160.10.1529. PMID 10826469
- [Result] Jimenez D, Aujesky D, Moores L, Gomez V, Lobo JL, Uresandi F, Otero R, Monreal M, Muriel A, Yusen RD; RIETE Investigators. Simplification of the pulmonary embolism severity index for prognostication in patients with acute symptomatic pulmonary embolism. Arch Intern Med. 2010 Aug 9;170(15):1383-9. doi: 10.1001/archinternmed.2010.199. PMID 20696966
- [Result] Elias A, Mallett S, Daoud-Elias M, Poggi JN, Clarke M. Prognostic models in acute pulmonary embolism: a systematic review and meta-analysis. BMJ Open. 2016 Apr 29;6(4):e010324. doi: 10.1136/bmjopen-2015-010324. PMID 27130162
- [Result] Agnelli G, Becattini C. Acute pulmonary embolism. N Engl J Med. 2010 Jul 15;363(3):266-74. doi: 10.1056/NEJMra0907731. Epub 2010 Jun 30. No abstract available. PMID 20592294
- [Result] Yu S, Zhou H, Li Y, Song J, Shao J, Wang X, Xie Z, Qiu C, Sun K. PERFORM: Pulmonary embolism risk score for mortality in computed tomographic pulmonary angiography-confirmed patients. EClinicalMedicine. 2021 May 31;36:100897. doi: 10.1016/j.eclinm.2021.100897. eCollection 2021 Jun. PMID 34136775